CLINICAL TRIAL: NCT04245670
Title: 5 Fractions of Pelvic SABR With Intra Prostatic SABR Boost:A Phase II Study (5STAR-PC)
Brief Title: 5 Fractions of Pelvic SABR With Intra Prostatic SABR Boost:
Acronym: 5STAR-PC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Prostate Cure Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5STAR-PC
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Ablative Body Radiotherapy (SABR) 35-50 Gy/5 (Experimental): Stereotactic Ablative Body Radiotherapy (SABR) given in 5 weekly fractions. Simultaneously treating the pelvic lymph nodes, prostate and MRI-nodule to a total dose of 25 Gy, 35 Gy and up to 50 Gy, respectively. The radiation will be given with 6-18 months of ADT.
  Interventions: Radiation: Stereotactic Ablative Body Radiotherapy (SABR) 35-50 Gy/5

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiotherapy (SABR) 35-50 Gy/5 — Stereotactic Ablative Body Radiotherapy (SABR) given in 5 weekly fractions. Simultaneously treating the pelvic lymph nodes, prostate and MRI-nodule to a total dose of 25 Gy, 35 Gy and up to 50 Gy, respectively. The radiation will be given with 6-18 months of ADT.

SUMMARY:
Stereotactic Ablative Body Radiotherapy (SABR) given in 5 weekly fractions. Simultaneously treating the pelvic lymph nodes, prostate and MRI-nodule to a total dose of 25 Gy, 35 Gy and up to 50 Gy, respectively. The radiation will be given with 6-18 months of ADT.

5-fraction SABR is a feasible, well-tolerated, effective and cost effective treatment for high-intermediate and high risk prostate cancer with/without an image-guided intraprostatic boost.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed prostate adenocarcinoma (centrally reviewed)
* High-intermediate risk defined as two or more of: T2c, Gleason 7 OR PSA 10-20ng/ml,
* High-risk prostate cancer, defined as at least one of: T3, Gleason 8-10, OR PSA > 20 ng/mL
* Willing to give informed consent to participate in this clinical trial
* Able and willing to complete EPIC, PORPUS and EQ-5D questionnaires

Exclusion Criteria

* Prior pelvic radiotherapy
* Contraindication to radical prostate radiotherapy e.g. connective tissue disease or inflammatory bowel disease
* Anticoagulation medication (if unsafe to discontinue for fiducial insertion)
* Diagnosis of bleeding diathesis
* Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >20
* Evidence of castrate resistance (defined as PSA < 3 ng/ml while testosterone is < 0.7nmol/l. Patients could have been on combined androgen blockade but are excluded if this was started due to PSA progression.
* Definitive extrapelvic nodal or distant metastatic disease on staging investigations.
* Hip prosthesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with Prostate cancer
Enrollment: 75 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity | Baseline to 3 months post completion of treatment
  To document the acute urinary toxicity using the Common Terminology Criteria for Adverse Events (CTCAE v4.0) criteria
Acute Toxicity | Baseline to 3 months post completion of treatment
  To document the acute bowel toxicity using the Common Terminology Criteria for Adverse Events (CTCAE v4.0) criteria

SECONDARY OUTCOMES:
Quality of Life outcome | Baseline to end of 5 year follow up
  Measuring quality of life using Expanded Prostate Index Composite (EPIC)
Biochemical disease-free survival | Baseline to end of 5 year follow up
  Biochemical disease-free survival
Quality of life outcome | Baseline to end of 5 year follow up
  Health utilities using the EQ-5D Quality of Life Questionnaire tool
Quality of life outcome | Baseline to end of 5 year follow up
  Health utilities using PORPUS-U Quality of Life Questionnaire tool
Economic analysis | Baseline to end of 5 year follow up
  Cost effectiveness of treatment.Quality of life and cost estimates will be captured for each patient from time of the initiation of treatment until death. The effectiveness endpoints will be biochemical disease free survival and quality-adjusted life years (QALYs). QALY will be calculated by survival (in years) multiplied by a utility weight associated with a certain condition.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontairo, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: Analysis of acute toxicity will be performed approximately 6 months after the last patient has been accrued, in August 2020. The final analysis will be performed when all patients have completed 5 years of follow-up, in early 2025.
Access Criteria: The primary endpoint analysis will be shared thru publications